CLINICAL TRIAL: NCT01375361
Title: Nebulized Albuterol for Congestive Heart Failure Exacerbation
Acronym: ACHE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RandomizedAlbuterolCHF
Record Dates: First submitted 2010-04-20; First posted 2011-06-17 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Congestive Heart Failure
Keywords: albuterol
MeSH Terms: conditions — Heart Failure | interventions — Albuterol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Albuterol (Experimental): Patients identified to have Cardiogenic Pulmonary Edema, will receive 2.5mg of Albuterol nebulizer on enrollment in the study and again at 4 hours. Patients will be monitored on telemetry in the emergency department during and after study drug administration. Although study drug administration will cease after 4 hours, we will continue to record ongoing data during the patient's hospitalization.
  Interventions: Drug: Albuterol
- Inhaled Placebo. (Placebo Comparator): Patients identified to have Cardiogenic Pulmonary Edema will receive 2.5mg Normal saline inhaled (Placebo) on enrollment and at 4 hours in the emergency department. Patient will be monitor on telemetry in the emergency department during and after placebo administration.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Albuterol — 2.5mg Albuterol inhaled on enrollment and at 4 hours in the emergency department.
  Other Names: Administration of Albuterol.
  Arms: Inhaled Albuterol
Drug: Normal Saline — 2.5mg Normal Saline inhaled on enrollment and at 4 hours in emergency department.
  Other Names: Administration of Placebo.
  Arms: Inhaled Placebo.

SUMMARY:
This is a randomized trial of the use of Albuterol in the setting of acute decompensated Congestive Heart Failure with radiographic evidence of Cardiogenic Pulmonary Edema.

DETAILED DESCRIPTION:
The objective is to carry out a randomized blinded placebo-controlled trial of inhaled Albuterol as an early therapy for patients with decompensated Congestive Heart Failure. Compared to placebo, inhaled Albuterol will improve oxygenation and decrease the need for non-invasive ventilation in patients with Cardiogenic Pulmonary Edema.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 with shortness of breath and history of CHF
* pulmonary edema on chest xr

Exclusion Criteria:

* pregnancy
* clinical or ekg changes to suggest acute coronary syndrome
* history of copd or asthma
* history of albuterol on medication list

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Borg Dyspnea Score | 8 hours.
  Patients are evaluated for approximatly 8 hours with the Borg Dyspnea Score. Starting at the time of arrival, then one hour later and consequently every two hours until reaching 8 hours in total.
  The Borg score is used to quantify the degree of shortness of breath a person is experiencing which is a measured on a 10 point visual-analog scale.

SECONDARY OUTCOMES:
Admission | An average of 48 hours
  If the patient is hospitalized we will continue to record information about their hospital stay and the patient will not receive more study interventions.

CONTACTS AND LOCATIONS:
Overall Officials: John C. Stein, MD., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States